CLINICAL TRIAL: NCT04575064
Title: An International Randomized Trial of Additional Treatments for COVID-19 in Hospitalized Patients Who Are All Receiving the Local Standard of Care - WHO-SOLIDARITY-GERMANY
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Explanation will be submitted later.
Sponsor: Professor Dr. Bernd Mühlbauer (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); World Health Organization (Other)
Responsible Party: Sponsor-Investigator, Professor Dr. Bernd Mühlbauer, Professor of Pharmacology - Head of Department, Klinikum Bremen-Mitte, gGmbH
Organization: Klinikum Bremen-Mitte, gGmbH (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WHO-SOLIDARITY-GERMANY; 2020-001549-38 (EudraCT Number)
Record Dates: First submitted 2020-09-30; First posted 2020-10-05 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: SARS-CoV-2 Infection; COVID-19; Moderate and Severe COVID-19
MeSH Terms: conditions — COVID-19; Lymphoma, Follicular | interventions — Standard of Care; remdesivir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SoC) (Other): This arm will receive standard supportive care according to guidelines for COVID-19. This is expected to vary regionally and may change throughout the trial based on new and emerging data on best care guidelines for patients.
  Interventions: Other: Standard of Care (SoC)
- Remdesivir + SoC (Experimental): Remdesivir 200 mg IV on day 1, followed by 100 mg IV daily infusion for 9 days plus optimized supportive care
  Interventions: Other: Standard of Care (SoC); Drug: Remdesivir

INTERVENTIONS:
Other: Standard of Care (SoC) — Standard supportive care is expected to vary regionally and may change throughout the trial based on new and emerging data on best care guidelines for patients.
Drug: Remdesivir — Remdesivir 200mg IV on day 1, followed by 100 mg IV daily infusion for 9 days or until discharge from hospital, whichever occurs first
  Arms: Remdesivir + SoC

SUMMARY:
This study is an adaptive, randomized, open-label, controlled clinical trial, performed worldwide in collaboration with WHO and INSERM.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Current SARS-CoV-2 infection
* Admitted to the hospital ward or the ICU due to COVID-19
* SpO2 <= 94% on room air OR oxygen demand OR breathing support
* Written informed consent obtained

Exclusion Criteria:

* Patient's non-consent or inability to informed consent
* Pregnant or breastfeeding women.
* Subjects pretreated with one of the study drugs in the past 29 days
* Anticipated transfer within 72 hours to a non-study hospital
* Severe co-morbidity with life expectancy < 3 months
* AST or ALT > 5 times the upper limit of normal
* Stage 4 severe chronic kidney disease or requiring dialysis
* Contraindications and known intolerance to any of the study drugs
* Subjects participating in a potentially confounding drug or device trial
* Any reason why the patient should not participate (investigator's opinion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Improvement of clinical status on the ordinal 7-point severity-scale at day 15. | at day 15
  WHO 7-point ordinal scale:
  1. Not hospitalized, no limitations on activities;
  2. Not hospitalized, limitation on activities;
  3. Hospitalized, not requiring supplemental oxygen;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  6. Hospitalized, on invasive mechanical ventilation or ECMO;
  7. Death

SECONDARY OUTCOMES:
Time to an improvement of one category from admission using the 7-point ordinal scale | up to 29 days
Mortality: 28 days mortality; in-house mortality | up to 29 days
Hospital stay: Duration of hospital stay due to COVID-19 | up to 29 days
Oxygen: Need of, time to first receiving and duration of oxygen | up to 29 days
Intensive care: Need of, time to first receiving and duration of intensive care | up to 29 days
Mechanical ventilation: Need of, time to first receiving and duration of mechanical ventilation | up to 29 days
ECMO: Need of, time to first receiving and duration for extracorporeal membrane oxygenation | up to 29 days
Superinfections, assessed with pathogen testing | up to 29 days
Kidney failure | up to 29 days
Myocardial failure | up to 29 days
Multiple organ failure | up to 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Welte, MD, Prof., Principal Investigator — Hannover Medical School
Locations (4):
- Germany (4):
  - Gesundheit Nord gGmbH, Bremen
  - Universitätsklinikum Gießen, Giessen
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Technische Universität München (TUM), München